CLINICAL TRIAL: NCT00903409
Title: OM6X: An Open-Label Extension of a Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Combined Lovaza (Previously Omacor®) and Simvastatin Therapy in Hypertriglyceridemic Subjects
Brief Title: Open-Label Extension of a Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Lovaza® and Simvastatin Therapy in Hypertriglyceridemic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 111818; LOV111858 (Other: GSK)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Hypertriglyceridemia
Keywords: High triglycerides; Lovaza; simvastatin; omega-3-acid ethyl esters
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Simvastatin; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin + Lovaza® ("Non-switchers") (Experimental): Open label Simvastatin + Lovaza® (omega-3-acid ethyl esters) NOTE: this group was originally assigned to Simvastatin + Lovaza® in the double-blind trial, hence in this open-label extension, they are termed "Non-switchers"
  Interventions: Drug: Simvastatin + Lovaza® (omega-3-acid ethyl esters)
- Simvastatin + Lovaza® ("Switchers") (Experimental): Open label Simvastatin + Lovaza® (omega-3-acid ethyl esters) NOTE: this group was originally assigned to Simvastatin + placebo in the double-blind trial, hence in this open-label extension, they are termed "Switchers"
  Interventions: Drug: Simvastatin + Lovaza® (omega-3-acid ethyl esters)

INTERVENTIONS:
Drug: Simvastatin + Lovaza® (omega-3-acid ethyl esters) — Open-label Simvastatin + Lovaza® (omega-3-acid ethyl esters) [formerly known as Omacor]

SUMMARY:
In a previous trial (LOV111858/OM6), subjects received in a double-blind fashion either 4 g/day of Lovaza® (omega-3-ethyl esters) [formerly known as Omacor] co-administered with simvastatin 40 mg/day or placebo co-administered with simvastatin 40 mg/day for 8 weeks. This extension trial, LOV111818/OM6X assessed the continued efficacy and safety of Lovaza® (omega-3-ethyl esters) co-administered with simvastatin 40 mg vs. switching from simvastatin plus placebo to simvastatin plus Lovaza® for lowering non-High Density Lipoprotein-Cholesterol (non-HDL-C) levels at 4 months (primary endpoint) and additionally at 12 and 24 months.

DETAILED DESCRIPTION:
Two studies comprise this OM6 Program. Study LOV111858/OM6 (double-blind study) which is outlined in NCT00246701 and Study LOV111818/OM6X (open-label extension) outlined in this posting.

ELIGIBILITY:
For LOV111818/OM6X - Subjects were included in the study if they had met all relevant inclusion/exclusion criteria prior to and throughout the double-blind Study LOV111858/OM6 and completed Study LOV111858/OM6 to Week 8.

FYI - entry criteria for LOV111818/OM6 (double-blind study)

Inclusion Criteria:

* Men and women ages 18-79 years, inclusive
* Current therapy with a statin drug
* Triglyceride levels between 200 and 499 mg/dL
* Normally active and in good health on the basis of medical history, brief physical examination, electrocardiogram, and routine laboratory tests
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Sensitivity to statin drugs or omega-3 fatty acids
* Lipoprotein lipase impairment or apo C-2 deficiency or type III hyperlipidemia
* Unexplained muscle pain or weakness
* History of pancreatitis
* Recent history of certain heart, kidney, liver, lung, or gastrointestinal diseases, or cancer (except non-melanoma skin cancer)
* Poorly controlled diabetes, or receiving insulin therapy
* Pregnant or lactating females. Women of childbearing potential who are not using a medically approved method of contraception.
* Use of certain types of hormones, anticonvulsant drugs, immunologic drugs, antibiotic, antifungal and antiviral drugs, and cardiac drugs
* Use of warfarin (Coumadin)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2005-11-15 (Actual); Primary Completion 2008-06-27 (Actual); Study Completion 2008-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (38):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Thousand Oaks, California
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Dunwoody, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Bloomington, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Wentzville, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Lakewood, Washington
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bays HE, Maki KC, McKenney J, Snipes R, Meadowcroft A, Schroyer R, Doyle RT, Stein E. Long-term up to 24-month efficacy and safety of concomitant prescription omega-3-acid ethyl esters and simvastatin in hypertriglyceridemic patients. Curr Med Res Opin. 2010 Apr;26(4):907-15. doi: 10.1185/03007991003645318. PMID 20156032
- [Background] Maki KC, Dicklin MR, Davidson MH, Doyle RT, Ballantyne CM; COMBination of prescription Omega-3 with Simvastatin (COMBOS) Investigators. Baseline lipoprotein lipids and low-density lipoprotein cholesterol response to prescription omega-3 acid ethyl ester added to Simvastatin therapy. Am J Cardiol. 2010 May 15;105(10):1409-12. doi: 10.1016/j.amjcard.2009.12.063. Epub 2010 Mar 30. PMID 20451686
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111818 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-switcher: Open-label Lovaza® (omega-3-acid ethyl esters) [formerly known as Omacor®] 4 g/day and Simvastatin 40 mg/day. These are the same drugs as administered in an earlier double-blind study (111858: NCT00903409).
- Switcher: Open-label Lovaza® (omega-3-acid ethyl esters) [formerly known as Omacor®] 4 g/day and Simvastatin 40 mg/day. Switched from Placebo/Simvastatin 40 mg/day administered in an earlier double-blind study (111858: NCT00903409).
Period: Overall Study
Arm/Group | Non-switcher | Switcher
Started | 88 | 100
Completed | 62 | 73
Not Completed | 26 | 27
Not completed — Adverse Event | 11 | 9
Not completed — Non-compliance with Protocol | 1 | 1
Not completed — Laboratory Abnormality | 2 | 0
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Other | 2 | 3
Not completed — Lost to Follow-up | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-switcher | Switcher | Total
Number analyzed (Participants) | 85 | 97 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.32) | 60.0 (10.80) | 59.9 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 49 | 59 | 108
Race/Ethnicity, Customized [Number; unit: Number of participants]
  White | 80 | 95 | 175
  Asian | 2 | 0 | 2
  Black or African American | 2 | 1 | 3
  Hispanic or Latino | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change of Non-HDL-C (High Density Lipoprotein-Cholesterol) in Switchers vs. Non-Switchers Subjects From LOV111858 End-of-Treatment (Week 8) to Month 4 of Extension Study (LOV111818)
Description: Median percent change from LOV111858 (NCT00903409) End-of-Treatment (double-blind study, Week 8) to the Month 4 visit of LOV111818 (open-label extension trial)
Time Frame: Month 4 (LOV111818)
Population: Intent-to-Treat (ITT) Population: Comprised of data for all participants who were enrolled and received at least one dose of study medication
Measure: Median (Full Range); unit: Percent change
Groups:
- Total Non-switcher and Switcher: Non-switcher and Switcher groups combined
Arm/Group | Non-switcher | Switcher | Total Non-switcher and Switcher
Number analyzed (Participants) | 80 | 92 | 172
Percent change | 0.9 [-47.5 to 60] | -9.4 [-35.7 to 33.9] | -3.3 [-47.5 to 60.0]
Statistical Analysis 1: Comparison: Non-switcher vs Switcher; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis — The difference between Non-switchers and Switchers in the percent change in non-HDL-C level from the end of the OM6 double-blind study (average of Weeks 6 and 8 for the statistical analysis) to 4 months of OM6X open-label treatment (Month 4)

2. Secondary Outcome: Median Percent Change of Lipid Measurements From LOV111858 End-of-Treatment Week 8 to Months 4, 12, and 24 of the Open-Label Extension Study (LOV111818) in "Switchers" vs. Non-switchers
Description: Median percent change from LOV111858 Baseline to LOV111818 Months 4, 12, and 24 visits of the open-label extension trial
Time Frame: Months 4, 12, and 24 (LOV111818) of the open-label extension trial
Population: ITT Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | Non-switcher | Switcher | Total Non-switcher and Switcher
Number analyzed (Participants) | 85 | 96 | 181
Percent change
  Non-HDL-C, Month 4 | -5.4 [-52.1 to 43.8] | -10.3 [-38.7 to 53.8] | -8.3 [-52.1 to 53.8]
  Non-HDL-C, Month 12 | -6.6 [-51.9 to 115.6] | -8.1 [-58.6 to 39.4] | -7.3 [-58.6 to 115.6]
  Non-HDL-C, Month 24 | -7.8 [-47.0 to 97.4] | -9.0 [-43.4 to 39.4] | -8.9 [-47.0 to 97.4]
  Triglycerides (TG), Month 4 | -26.2 [-71.0 to 130.5] | -31.5 [-64.6 to 59.7] | -29.8 [-71.0 to 130.5]
  TG, Month 12 | -30.4 [-75.9 to 189.6] | -35.7 [-71.8 to 59.7] | -34.6 [-75.9 to 189.6]
  TG, Month 24 | -28.2 [-86.1 to 138.7] | -35.7 [-74.5 to 59.7] | -33.3 [-86.1 to 138.7]
  Total-Cholesterol (Total-C), Month 4 | -4.2 [-41.6 to 32.3] | -7.7 [-27.7 to 46.9] | -6.5 [-41.6 to 46.9]
  Total-C, Month 12 | -5.4 [-31.5 to 83.9] | -7.7 [-52.6 to 34.6] | -6.5 [-52.6 to 83.9]
  Total-C, Month 24 | -6.4 [-40.6 to 69.6] | -6.8 [-32.2 to 34.6] | -6.7 [-40.6 to 69.6]
  Calculated Very Low Density (VLD)L-C, Month 4 | -24.3 [-65.2 to 86.4] | -29.3 [-64.6 to 47.6] | -27.9 [-65.2 to 86.4]
  Calculated Very Low Density (VLD)L-C, Month 12 | -29.8 [-75.8 to 62.2] | -31.9 [-71.8 to 45.2] | -30.7 [-75.8 to 62.2]
  Calculated Very Low Density (VLD)L-C, Month 24 | -25.0 [-68.8 to 213.6] | -33.1 [-74.1 to 45.2] | -31.5 [-74.1 to 213.6]
  Low Density (LD)L-C, Month 4 | 2.4 [-38.4 to 77.4] | -0.4 [-30.3 to 88.1] | 1.7 [-38.4 to 88.1]
  Low Density (LD)L-C, Month 12 | 5.9 [-34.6 to 73.4] | 6.3 [-33.8 to 63.4] | 6.2 [-34.6 to 73.4]
  Low Density (LD)L-C, Month 24 | 3.4 [-34.1 to 186.2] | 2.6 [-32.0 to 70.9] | 3.0 [-34.1 to 186.2]
  HDL-C, Month 4 | 0.8 [-29.4 to 39.8] | 0.0 [-22.2 to 31.9] | 0.0 [-29.4 to 39.8]
  HDL-C, Month 12 | 0.0 [-33.3 to 50.0] | -3.1 [-23.2 to 44.1] | -0.9 [-33.3 to 50.0]
  HDL-C, Month 24 | -2.9 [-44.8 to 50.0] | -5.6 [-37.7 to 36.0] | -4.6 [-44.8 to 50.0]
  Total-C:HDL-C Ratio, Month 4 | -5.3 [-39.6 to 78.0] | -7.9 [-35.8 to 30.2] | -6.9 [-39.6 to 78.0]
  Total-C:HDL-C Ratio, Month 12 | -3.6 [-39.6 to 139.5] | -4.7 [-38.3 to 42.2] | -4.0 [-39.6 to 139.5]
  Total-C:HDL-C Ratio, Month 24 | -1.9 [-39.3 to 154.9] | -3.8 [-44.5 to 60.8] | -3.5 [-44.5 to 154.9]

3. Secondary Outcome: Median Percent Change of Lipid Measurements From LOV111858 End-of-Treatment Week 8 to LOV111818 Months 4, 12, and 24 of the Open-Label Extension Trial
Description: Median percent change from LOV111858 End-of-Treatment (Week 8) to LOV111818 Months 4, 12, and 24 visits of the open-label extension trial
Time Frame: LOV111858 End-of-Treatment (Week 8) to LOV111818 Months 4, 12, and 24 of the open-label extension trial
Population: ITT Population
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Non-switcher | Switcher | Total Non-switcher and Switcher
Number analyzed (Participants) | 85 | 96 | 181
Percentage change
  Non-HDL-C, Month 12 | -0.2 [-44.1 to 76.7] | -6.4 [-58.6 to 29.2] | -1.5 [-58.6 to 76.7]
  Non-HDL-C, Month 24 | 1.6 [-39.0 to 102.8] | -6.3 [-35.0 to 40.7] | -3.8 [-39.0 to 102.8]
  TG Month, 4 | 1.8 [-52.1 to 134.1] | -25.8 [-69.5 to 39.4] | -15.8 [-69.5 to 134.1]
  TG Month, 12 | -3.2 [-58.6 to 194.2] | -27.0 [-71.8 to 97.2] | -17.1 [-71.8 to 194.2]
  TG Month, 24 | -6.4 [-81.2 to 390.1] | -27.0 [-74.7 to 97.2] | -19.5 [-81.2 to 390.1]
  Total-C, Month 4 | 0.6 [-37.7 to 40.4] | -7.1 [-29.3 to 25.3] | -2.5 [-37.7 to 40.4]
  Total-C, Month 12 | -1.7 [-23.2 to 58.9] | -3.4 [-53.2 to 23.9] | -2.7 [-53.2 to 58.9]
  Total-C, Month 24 | -1.0 [-30.2 to 53.5] | -5.6 [-31.1 to 34.2] | -3.0 [-31.1 to 53.5]
  Calculated VLDL-C, Month 4 | 2.1 [-52.9 to 122.7] | -23.1 [-69.2 to 38.0] | -13.5 [-69.2 to 122.7]
  Calculated VLDL-C, Month 12 | -4.6 [-58.6 to 113.6] | -21.3 [-69.8 to 97.2] | -13.7 [-69.8 to 113.6]
  Calculated VLDL-C, Month 24 | -5.8 [-80.7 to 113.6] | -26.4 [-71.1 to 97.2] | -17.5 [-80.7 to 113.6]
  LDL-C, Month 4 | 0.6 [-45.7 to 64.3] | 6.3 [-35.4 to 56.7] | 3.7 [-45.7 to 64.3]
  LDL-C, Month 12 | 1.9 [-28.2 to 64.7] | 10.1 [-32.1 to 69.8] | 6.3 [-32.1 to 69.8]
  LDL-C, Month 24 | 1.9 [-28.6 to 105.9] | 5.5 [-32.2 to 80.1] | 3.8 [-32.2 to 105.9]
  HDL-C, Month 4 | -2.9 [-33.3 to 31.1] | 1.7 [-22.8 to 34.8] | -1.2 [-33.3 to 34.8]
  HDL-C, Month 12 | -3.1 [-34.1 to 30.8] | -1.8 [-30.7 to 40.4] | -2.8 [-34.1 to 40.4]
  HDL-C, Month 24 | -5.4 [-41.8 to 30.8] | -4.8 [-40.6 to 21.9] | -4.9 [-41.8 to 30.8]
  Total-C:HDL-C Ratio, Month 4 | 1.3 [-33.4 to 110.5] | -7.5 [-31.8 to 35.5] | -3.5 [-33.4 to 110.5]
  Total-C:HDL-C Ratio, Month 12 | 2.7 [-35.5 to 96.1] | -5.4 [-34.9 to 53.4] | -0.1 [-35.5 to 96.1]
  Total-C:HDL-C Ratio, Month 24 | 5.7 [-36.7 to 116.3] | -1.9 [-31.4 to 58.8] | 1.1 [-36.7 to 116.3]

ADVERSE EVENTS:
Arm/Group | Non-switcher | Switcher | Total Non-switcher and Switcher
Serious Adverse Events (participants affected / at risk) | 17 | 11 | 28
Other Adverse Events (participants affected / at risk) | 67 | 79 | 146
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Non-switcher | Switcher | Total Non-switcher and Switcher
Atrial fibrillation (Cardiac disorders) | 2/85 | 0/97 | 2/182
Coronary artery disease (Cardiac disorders) | 2/85 | 0/97 | 2/182
Myocardial infarction (Cardiac disorders) | 0/85 | 2/97 | 2/182
Acute myocardial infarction (Cardiac disorders) | 1/85 | 0/97 | 1/182
Aortic valve stenosis (Cardiac disorders) | 0/85 | 1/97 | 1/182
Pericardial infusion (Cardiac disorders) | 1/85 | 0/97 | 1/182
Back pain (Musculoskeletal and connective tissue disorders) | 1/85 | 0/97 | 1/182
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0/85 | 1/97 | 1/182
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/85 | 0/97 | 1/182
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0/85 | 1/97 | 1/182
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/85 | 1/97 | 1/182
Cellulitis (Infections and infestations) | 1/85 | 0/97 | 1/182
Gastroenteritis (Infections and infestations) | 0/85 | 1/97 | 1/182
Pneumonia (Infections and infestations) | 0/85 | 1/97 | 1/182
Pancreatitis (Gastrointestinal disorders) | 1/85 | 0/97 | 1/182
Small Intestinal Obstruction (Gastrointestinal disorders) | 1/85 | 0/97 | 1/182
Femoral neck fracture (Injury, poisoning and procedural complications) | 1/85 | 0/97 | 1/182
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1/85 | 0/97 | 1/182
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/85 | 0/97 | 1/182
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/85 | 0/97 | 1/182
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/85 | 0/97 | 1/182
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/85 | 1/97 | 1/182
Hyperparathyroidism (Endocrine disorders) | 1/85 | 0/97 | 1/182
Chest discomfort (General disorders) | 1/85 | 0/97 | 1/182
Hepatic steatosis (Hepatobiliary disorders) | 0/85 | 1/97 | 1/182
Dehydration (Metabolism and nutrition disorders) | 1/85 | 0/97 | 1/182
Carotid artery occlusion (Nervous system disorders) | 0/85 | 1/97 | 1/182
Bipolar disorder (Psychiatric disorders) | 1/85 | 0/97 | 1/182
Nephrolithiasis (Renal and urinary disorders) | 1/85 | 0/97 | 1/182
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/85 | 0/97 | 1/182
Deep vein thrombosis (Vascular disorders) | 0/85 | 1/97 | 1/182
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Non-switcher | Switcher | Total Non-switcher and Switcher
Hypertension (Vascular disorders) | 7/85 | 13/97 | 20/182
Bronchitis (Infections and infestations) | 5/85 | 10/97 | 15/182
Sinusitis (Infections and infestations) | 9/85 | 5/97 | 14/182
Arthralgia (Musculoskeletal and connective tissue disorders) | 6/85 | 6/97 | 12/182
Upper respiratory tract infection (Infections and infestations) | 5/85 | 7/97 | 12/182
Nasopharyngitis (Infections and infestations) | 5/85 | 5/97 | 10/182
Diarrhea (Gastrointestinal disorders) | 2/85 | 7/97 | 9/182
Myalgia (Musculoskeletal and connective tissue disorders) | 6/85 | 3/97 | 9/182
Urinary tract infection (Infections and infestations) | 3/85 | 6/97 | 9/182
Anxiety (Psychiatric disorders) | 5/85 | 3/97 | 8/182
Back pain (Musculoskeletal and connective tissue disorders) | 3/85 | 5/97 | 8/182
Dyspepsia (Gastrointestinal disorders) | 5/85 | 2/97 | 7/182
Depression (Psychiatric disorders) | 5/85 | 2/97 | 7/182
Weight increased (Investigations) | 1/85 | 5/97 | 6/182

LIMITATIONS AND CAVEATS:
Only Adverse Experience categories with a greater than 5% occurrence in any group were reported in the AE table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.